CLINICAL TRIAL: NCT06018701
Title: A Clinical Trial of Dental Device Made of Zirconia Cemented with PMMA Bone Cement on Partial Edentulous Patients of Kathmandu
Brief Title: A Clinical Trial of Dental Device Cemented with Polymethyl Methacrylate (PMMA) Bone Cement
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bluebird International Clinic (Other)
Responsible Party: Principal Investigator, Parakram Parajuli, Principal Investigator, Bluebird International Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BluebirdIC
Record Dates: First submitted 2023-07-26; First posted 2023-08-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Edentulism

STUDY DESIGN:
Intervention Model Description: Total forty eight (48) dental devices made of zirconia will be cemented. 12 dental device in each allocated quadrant, i.e., maxillary anterior, maxillary posterior, mandibular anterior and mandibular posterior. And the results will be compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Maxillary Anterior (Experimental): Dental device will be cemented with PMMA bone cement on group that have missing tooth on maxillary anterior region.
  Interventions: Device: A dental device made of zirconia. This is a new invention and does not exist generically. The given generic name of the invention (dental device) is "Dantya Nikhan".
- Maxillary Posterior (Experimental): Dental device will be cemented with PMMA bone cement on group that have missing tooth on maxillary posterior region.
  Interventions: Device: A dental device made of zirconia. This is a new invention and does not exist generically. The given generic name of the invention (dental device) is "Dantya Nikhan".
- Mandibular Anterior (Experimental): Dental device will be cemented with PMMA bone cement on group that have missing tooth on mandibular anterior region.
  Interventions: Device: A dental device made of zirconia. This is a new invention and does not exist generically. The given generic name of the invention (dental device) is "Dantya Nikhan".
- Mandibular Posterior (Experimental): Dental device will be cemented with PMMA bone cement on group that have missing tooth on mandibular posterior region.
  Interventions: Device: A dental device made of zirconia. This is a new invention and does not exist generically. The given generic name of the invention (dental device) is "Dantya Nikhan".

INTERVENTIONS:
Device: A dental device made of zirconia. This is a new invention and does not exist generically. The given generic name of the invention (dental device) is "Dantya Nikhan". — Dental device is surgically placed and cemented with PMMA bone cement on edentulous region.
  Other Names: "Dantya Nikhan" is a generic given "Sanskrit" name, as it is a new invention and does not currently exist publicly.

SUMMARY:
Conventional bridge and dental implants have been playing a significant role in replacing missing tooth/teeth. But they come with shortcomings. Hence, to explore the possibility of addressing such shortcomings, a clinical trial study of a new dental device made of zirconia is intended to be studied to see if it could serve as an additional option for fixed prosthodontics. An approach to explore possibilities for cheaper and faster procedure with regards to the treatment of tooth/teeth loss.

DETAILED DESCRIPTION:
Objectives:

To determine whether the use of a new dental device made of zirconia cemented with Polymethyl methacrylate (PMMA) bone cement could be an additional option for a faster treatment for missing tooth/teeth with fixed/removable prosthodontics.

Methodology:

After a Cone Beam Computed Tomography (CBCT) scan and clinical evaluation, 48 samples of zirconia dental device will be cemented with PMMA bone cement in edentulous area on randomized population. Immediate loading (0-15 days) with single crown and multiple unit bridge made of zirconia will be cemented using luting cement as fixed restoration. Radiographic evaluation and clinical examination will be conducted every three (3) months for one year.

Expected Outcome:

A new dental device made of zirconia could be an additional option for the treatment of edentulism, which could be completed within 0-15 days with minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old and above) who agrees for the treatment
* Single/multiple missing tooth/teeth (edentulism)
* Maxillary/mandibular bone density of more than 350 Hounsfield Unit (HU)
* Edentulous region with minimum of 2mm bone width and 5mm of bone height
* Well controlled diabetes and hypertension

Exclusion Criteria:

* Severe/Critical medical conditions
* Adults above 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss around dental device ("dantya nikhan") measured in millimeters (mm) through intra-oral x-ray and horizontal and vertical bone loss through Cone Beam Computed Tomography (CBCT) Scan | Total time frame is 16 months, 48 samples trial is to be completed in 4 months. Each sample will have follow up of 3 months for 12 months. The trial of samples on 4th month will complete the 12 months follow up in the 16th month.
  During each visit of the participant every three (3) months (four times in twelve months), or as requested by the participant, intra-oral x-ray will be taken to evaluate hard tissue. Marginal bone loss, if any will be recorded in millimeters (mm). If additional issue (specially radiolucency) of hard tissue is detected then further evaluation through Cone Beam Computed Tomography (CBCT) Scan will be conducted.
Gingival status and health around dental device ("dantya nikhan") measured through Loe and Silness Gingival Index as Grade 0 to 3 and will be recorded with photographs | Total time frame is 16 months, 48 samples trial is to be completed in 4 months. Each sample will have follow up of 3 months for 12 months. The trial of samples on 4th month will complete the 12 months follow up in the 16th month.
  During each visit of the participant every three months (four times in twelve months), or as requested by the participant, clinical examination including photographs will be conducted to evaluate soft tissue. Additionally Loe and Silness Gingival Index will be used to measure in grades 0 to 3, where Grade 0 means Normal gingiva (natural coral pink gingiva; no inflammation; no discoloration); Grade 1 means Mild Inflammation (slight change in color; slight edema; no bleeding upon probing); Grade 2 means Moderate inflammation (Redness; edema; glazing; bleeding upon probing); and Grade 3 means Severe inflammation (Marked redness and edema; swelling; possible ulceration; tendency to bleed spontaneously).
Oral Hygiene status around dental device ("dantya nikhan") measured through Quigley and Hein Plaque Index as Score 0 to 5 | Total time frame is 16 months, 48 samples trial is to be completed in 4 months. Each sample will have follow up of 3 months for 12 months. The trial of samples on 4th month will complete the 12 months follow up in the 16th month.
  During each visit of the participant every three months (four times in twelve months), or as requested by the participant, Quigley and Hein Plaque Index will be used to evaluate oral hygiene through Score 0 to 5, where Score 0 means No Plaque; Score 1 means Flecks of stain on the gingival margin; Score 2 means Definite line of plaque on the gingival margin; Score 3 means Plaque on gingival third of tooth surface; Score 4 means Plaque on almost two thirds of tooth surface; and Score 5 means Plaque on greater than two third of tooth surface.
Pain on and around dental device ("dantya nikhan") measured through Visual Analogue Scale as Score 0 to 10 | Total time frame is 16 months, 48 samples trial is to be completed in 4 months. Each sample will have follow up of 3 months for 12 months. The trial of samples on 4th month will complete the 12 months follow up in the 16th month.
  During each visit of the participant every three months (four times in twelve months), or as requested by the participant, pain on and around dental device ("dantya nikhan") will be recorded with Visual Analogue Scale through Score 0 to 10, where Score 0 means No Pain; Score 1-3 means Mild Pain; Score 4-5 means Moderate Pain; Score 6-7 means Severe Pain; Score 8-9 means Very Severe Pain; and Score 10 means Worst Pain.
Discomfort on and around dental device ("dantya nikhan") measured through Visual Analogue Scale as Score 0 to 10 | Total time frame is 16 months, 48 samples trial is to be completed in 4 months. Each sample will have follow up of 3 months for 12 months. The trial of samples on 4th month will complete the 12 months follow up in the 16th month.
  During each visit of the participant every three months (four times in twelve months), or as requested by the participant, discomfort on and around dental device ("dantya nikhan") will be recorded with Visual Analogue Scale through Score 0 to 10, where Score 0 means No Discomfort; Score 1-3 means Mild Discomfort; Score 4-5 means Moderate Discomfort; Score 6-7 means Severe Discomfort; Score 8-9 means Very Severe Discomfort; and Score 10 means Worst Discomfort.
Dislodgment of dental device ("dantya nikhan") measured through Present, Mobile and Absent | Total time frame is 16 months, 48 samples trial is to be completed in 4 months. Each sample will have follow up of 3 months for 12 months. The trial of samples on 4th month will complete the 12 months follow up in the 16th month.
  During each visit of every three months (four times in twelve months), or as requested by the participant, dislodgment of dental device ("dantya nikhan") will be recorded through Present, Mobile and Absent, where Present means that the dental device has been completely detached from the osteotomy; Mobile means that the dental device is not completely detached, but is mobile; and Absent means that the dental device is neither completely detached from the osteotomy nor is mobile.
Fracture or crack of dental device ("dantya nikhan") measured through Present and Absent | Total time frame is 16 months, 48 samples trial is to be completed in 4 months. Each sample will have follow up of 3 months for 12 months. The trial of samples on 4th month will complete the 12 months follow up in the 16th month.
  During each visit every three months (four times in twelve months), or as requested by the participant, fracture of dental device ("dantya nikhan") will be recorded through Present and Absent, where Present means that the dental device is fractured or cracked; and Absent means that the dental device is neither fractured nor cracked.

CONTACTS AND LOCATIONS:
Overall Officials: Rabindra Mn Shrestha, MDS, Study Chair — Kantipur Dental College
Locations (1):
- Bluebird International Clinic, Kathmandu, Bagmati, Nepal